CLINICAL TRIAL: NCT01550302
Title: The Effect of Superficial Cervical Plexus Block on Post-Thoracotomy/Scopy Ipsilateral Shoulder Pain
Brief Title: Superficial Cervical Plexus Block for Shoulder Pain After Lung Surgery
Acronym: SCPB
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to continue enrollment due to lack of resources (research coordinator no longer available).
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Srdjan Jelacic, Assistant Professor, Anesthesiology & Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 42272
Record Dates: First submitted 2012-03-01; First posted 2012-03-09 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Shoulder Pain
Keywords: Superficial Cervical Plexus Block; Thoracic Surgery; Thoracotomy; Video-Assisted Thoracoscopic Surgery
MeSH Terms: conditions — Shoulder Pain | interventions — Cervical Plexus Block; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Controls (No Intervention): Subjects enrolled in this group will only have a line drawn on the side of their neck for superficial cervical plexus block, but we will not perform the injection. The subjects will not be aware whether they received an intra-operative block or not. In addition, neither the Post-Anesthesia Care Unit nurse nor the providers involved in the post-operative care will be aware of subjects group assignment.
- Superficial Cervical Plexus Block (Active Comparator): Subjects enrolled in this group will have a line drawn and will receive a superficial cervical plexus block at the end of the surgery just prior to emergence from anesthesia.
  Interventions: Procedure: Superficial Cervical Plexus Block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Superficial Cervical Plexus Block — At the end of the lung surgery while subjects are still under general anesthesia, one of the investigators will perform superficial cervical plexus. First, a line extending from the mastoid process to C6 transverse process is drawn. The site of needle insertion is marked at the midpoint of the line connecting the mastoid process with Chassaignac's tubercle of C6 transverse process. After skin cleansing with chlorhexidine prep, using a "fan" technique with superior-inferior needle redirections, 15 ml of 0.25% bupivacaine will be injected alongside the posterior border of the sternocleidomastoid muscle 2-3 cm below and above the needle insertion site.
  Other Names: Cervical Plexus Block
  Arms: Superficial Cervical Plexus Block
Drug: Bupivacaine — Single dose of 37.5 mg of bupivacaine subcutaneously
  Other Names: Marcain, Marcaine, Sensorcaine and Vivacaine
  Arms: Superficial Cervical Plexus Block

SUMMARY:
The investigators want to know whether injecting numbing medication on the side of the neck (also called superficial cervical plexus block) can prevent or reduce shoulder pain that patients commonly experience after lung surgery. The investigators will perform the injection at the end of your surgery while the subjects are still under general anesthesia and before they wake up. The investigators will use a local anesthetic (bupivacaine or Marcaine®) that is routinely used for skin infiltration of the surgical wounds.

This study is randomized and single-blind. This means that subjects will be assigned by chance (like flipping a coin) to receive either an injection with active medication (bupivacaine), or no injection at all.

DETAILED DESCRIPTION:
Pain management following lung surgery is of outmost importance. Providing adequate pain control facilitates patient recovery and improves lung function, therefore, leading to reduced morbidity and mortality associated with lung surgery. It is now well-established that lung surgery is associated with significant incisional pain, which in some patients may lead to development of chronic post-thoracotomy pain syndrome. In addition, many patients report significant shoulder pain that is often resistant to increasing epidural infusions and intravenous opioid therapy. The incidence of shoulder pain varies from study to study with estimates anywhere between 41% to 97%. Although the cause of the shoulder pain is not well understood, there are only few therapies available for the treatment of shoulder pain including acetaminophen, non-steroidal anti-inflammatory drugs, interscalene brachial plexus and stellate ganglion block. However, all of the currently available therapies have potentially significant side-effects. The investigators are not aware of any studies evaluating the effectiveness of superficial cervical plexus block in reducing or preventing shoulder pain following thoracotomy or thoracoscopic surgery. The superficial cervical plexus block is minimal risk procedure equivalent to an IV start.

The primary aim of this study is to compare the effect of superficial cervical plexus block when added to thoracic epidural analgesia and intravenous patient controlled analgesia (PCA) to standard thoracic epidural analgesia and PCA used at our institution on the incidence of shoulder pain.

Subjects participating in this study will receive standard clinical care in addition to the following research procedures:

* Intra-operative block: an injection of bupivacaine on the side of the neck at the end of the surgery while the subject is still under general anesthesia or no injection at all if in control group. If the subject is assigned to receive an injection, the investigators will be using a small needle similar to the one used to numb the skin for the IV start. There will be a single needle stick on the side of the neck (same side as the lung surgery) and injection of 15 mL of 0.25% bupivacaine under the skin. Regardless of whether the subject gets an injection or not, he/she will receive standard clinical care.
* Post-lung surgery pain assessment: the investigators will ask the subjects to rate their pain at the incision site, chest tube site and shoulder at rest and with movement at 6, 12, 18, 24 and 48 hours after lung surgery. The investigators will also ask the subjects about any side-effects that may be associated with the standard narcotic pain medications.

The investigators will collect the following data from the medical record including:

* Presence or absence of shoulder pain
* The amount of pain medicines (narcotics) needed to treat subject's pain over 24 and 48 hours after lung surgery
* The presence of any side-effects of narcotic pain medications
* Blood pressure, heart rate, EKG and oxygen levels when available in order to evaluate if improved shoulder pain and less narcotics used will have additional beneficial effects

Subjects are eligible if they are age 18-75 years and undergoing lung surgery.

Subjects are not eligible if they are non-English speaking, have had a previous lung surgery, are allergic to bupivacaine, have a history of chronic pain or have been taking pain medications for a long time, and already have shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* subjects who clinically consented to elective thoracotomy or video-assisted thoracoscopic surgery (VATS) under general anesthesia and epidural analgesia
* ages between 18 and 75 years

Exclusion Criteria:

* inability to perform thoracic epidural
* violation of protocol (e.g., administration of medication that does not comply with the study protocol)
* subject has change of mind
* surgery has to be repeated

Non-inclusion Criteria:

* subject refusal
* non-English speaking
* previous chronic or neuropathic pain
* previous chronic use of opioids
* history of psychiatric disorder
* allergy to local anesthetic
* previous ipsilateral thoracotomy or VATS
* prior history of shoulder pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan Jelacic, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] MacDougall P. Postthoracotomy shoulder pain: diagnosis and management. Curr Opin Anaesthesiol. 2008 Feb;21(1):12-5. doi: 10.1097/ACO.0b013e3282f2bb67. PMID 18195603
- [Background] Burgess FW, Anderson DM, Colonna D, Sborov MJ, Cavanaugh DG. Ipsilateral shoulder pain following thoracic surgery. Anesthesiology. 1993 Feb;78(2):365-8. doi: 10.1097/00000542-199302000-00023. No abstract available. PMID 8439033
- [Background] Pandit JJ, Dutta D, Morris JF. Spread of injectate with superficial cervical plexus block in humans: an anatomical study. Br J Anaesth. 2003 Nov;91(5):733-5. doi: 10.1093/bja/aeg250. PMID 14570798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Controls | Superficial Cervical Plexus Block
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls | Superficial Cervical Plexus Block | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (8.7) | 58.8 (6.7) | 58.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Height [Mean (Standard Deviation); unit: cm] | 181.0 (7.6) | 156.4 (4.6) | 168.7 (13.8)
Weight [Mean (Standard Deviation); unit: kg] | 89.7 (6.0) | 66.2 (18.7) | 77.9 (18.2)
Duration of Surgery [Mean (Standard Deviation); unit: minutes] | 181 (70) | 251 (108) | 216 (96)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-thoracotomy/Scopy Ipsilateral Shoulder Pain
Time Frame: 24 hours after lung surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Controls | Superficial Cervical Plexus Block
Number analyzed (Participants) | 5 | 5
Participants | 2 | 3

2. Secondary Outcome: Post-operative Opioid Consumption Expressed in Morphine Equivalents
Time Frame: 24 hours after the surgery
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Controls | Superficial Cervical Plexus Block
Number analyzed (Participants) | 5 | 5
mg | 30.0 (39.16) | 17.2 (17.5)

3. Secondary Outcome: Numeric Response Scale Pain Scores Around Ipsilateral Shoulder at Rest and During Movement
Description: Data collected on an interval scale ranging from 0 (no pain) to 10 (highest or most pain). Reported data shows an average of scores across participants
Time Frame: 6, 12, 18, 24 and 48 hours after the surgery
Population: Data not collected for 6, 12, and 18 hours at rest or with movement/coughing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls | Superficial Cervical Plexus Block
Number analyzed (Participants) | 5 | 5
units on a scale
  At rest 6 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 6 hrs: number analyzed (Participants) | 0 | 0
  At rest 12 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 12 hrs: number analyzed (Participants) | 0 | 0
  At rest 18 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 18 hrs: number analyzed (Participants) | 0 | 0
  At rest 24 hrs | 2.8 (4.21) | 4 (3.00)
  With movement 24 hrs | 2.8 (4.21) | 5.6 (3.13)
  At rest 48 hrs | 2.2 (3.03) | 4.6 (4.62)
  With movement 48 hrs | 3.4 (3.13) | 5.8 (4.38)

4. Secondary Outcome: Numeric Response Scale Pain Scores at Incision Site at Rest and During Coughing
Description: as for outcome 3
Time Frame: 6, 12, 18, 24 and 48 hours after the surgery
Population: Data not collected for 6, 12, and 18 hours at rest or moving/with cough
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls | Superficial Cervical Plexus Block
Number analyzed (Participants) | 5 | 5
units on a scale
  At rest 6 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 6 hrs: number analyzed (Participants) | 0 | 0
  At rest 12 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 12 hrs: number analyzed (Participants) | 0 | 0
  At rest 18 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 18 hrs: number analyzed (Participants) | 0 | 0
  At rest 24 hrs | 4.4 (4.04) | 3.2 (4.38)
  Movement or cough 24 hrs | 5.2 (4.15) | 7 (4.06)
  At rest 48 hrs | 1.6 (2.19) | 3.4 (4.67)
  Movement or cough 48 hrs | 3.8 (3.03) | 5.2 (4.15)

5. Secondary Outcome: Numeric Response Scale Pain Scores Around Chest Tube Insertion Site at Rest and During Coughing
Description: as for outcome 3
Time Frame: 6, 12, 18, 24 and 48 hours after the surgery
Population: Data not collected for 6, 12, and 18 hours at rest or with movement/cough
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls | Superficial Cervical Plexus Block
Number analyzed (Participants) | 5 | 5
units on a scale
  At rest 6 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 6 hrs: number analyzed (Participants) | 0 | 0
  At rest 12 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 12 hrs: number analyzed (Participants) | 0 | 0
  At rest 18 hrs: number analyzed (Participants) | 0 | 0
  Movement or cough 18 hrs: number analyzed (Participants) | 0 | 0
  At rest 24 hrs | 2.6 (2.88) | 5.8 (4.44)
  Movement or cough 24 hrs | 3.6 (3.58) | 7.2 (3.56)
  At rest 48 hrs | 1.6 (2.61) | 2.2 (2.59)
  Movement or cough 48 hrs | 4.2 (3.11) | 5.2 (3.70)

6. Secondary Outcome: Number of Participants Requiring Post-operative Ibuprofen as a Rescue Medication
Time Frame: 48 hours after the surgery
Measure: Number; unit: number of participants
Arm/Group | Controls | Superficial Cervical Plexus Block
Number analyzed (Participants) | 5 | 5
number of participants | 0 | 1

7. Secondary Outcome: Number of Patients With Post-operative Side Effects Such as Post-operative Nausea and Vomiting (PONV), Pruritus, Sedation, Respiratory Depression and Hypotension
Time Frame: 24 and 48 hours after the surgery
Population: Hypotension data not collected
Measure: Count of Participants; unit: Participants
Arm/Group | Controls | Superficial Cervical Plexus Block
Number analyzed (Participants) | 5 | 5
Participants
  PONV 24 hrs | 2 | 1
  PONV 48 hrs | 2 | 4
  Pruritis 24 hrs | 1 | 1
  Pruritis 48 hrs | 2 | 0
  Dizziness 24 hrs | 0 | 0
  Dizziness 48 hrs | 0 | 1
  Sedation 24 hrs | 1 | 0
  Sedation 48 hrs | 0 | 0
  Respiratory Depression 24 hrs | 1 | 0
  Respiratory Depression 48 hrs | 1 | 0
  Hypotension 24 hrs: number analyzed (Participants) | 0 | 0
  Hypotension 48 hrs: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Controls | Superficial Cervical Plexus Block
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No